CLINICAL TRIAL: NCT06875622
Title: Comparison of Behaviorally-Based Remote Approaches to Optimize Weight Loss and Identification of Factors Which Characterize Treatment Response
Brief Title: Remote Approaches for Optimizing Weight Loss (Elevate Weight Loss Trial)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2185718
Record Dates: First submitted 2025-03-08; First posted 2025-03-13 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Obesity/therapy
Keywords: behavioral weight loss; remote interventions; diet and exercise
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Automated online program + coaching (Experimental): Participants randomized to this condition will receive a 12-month automated weight loss program delivered via the Internet plus monthly, individual coaching sessions delivered via videoconference.
  Interventions: Behavioral: Automated online weight loss program; Behavioral: Individual coaching
- Automated online program only (Experimental): Participants randomized to this condition will receive a 12-month automated weight loss program delivered via the Internet.
  Interventions: Behavioral: Automated online weight loss program
- Group videoconference program + coaching (Experimental): Participants randomized to this condition will receive a 12-month, group-based behavioral weight loss program delivered via videoconference plus monthly, individual coaching sessions delivered via videoconference.
  Interventions: Behavioral: Individual coaching; Behavioral: Group-based, videoconference-delivered weight loss
- Group videoconference program only (Experimental): Participants randomized to this condition will receive a 12-month, group-based behavioral weight loss program delivered via videoconference.
  Interventions: Behavioral: Group-based, videoconference-delivered weight loss

INTERVENTIONS:
Behavioral: Automated online weight loss program — Participants receiving this program are given a daily calorie intake goal of 1200-1800 kcal/day based upon their starting weight and a moderate-intensity aerobic exercise (e.g., walking) goal which progresses to 250 min/week. They are instructed to self-monitor body weight, calorie intake, and exercise minutes daily over 12 months, and are provided with a smart scale for electronic transmission of weight data. Computer-generated, personalized feedback is based upon self-monitoring data, and provided weekly during months 1-3, twice per month during months 4-6, and monthly thereafter. Participants are also instructed to view a new multi-media video lesson weekly during months 1-3, 2x/month during months 4-6, and monthly thereafter (24 lessons in total). These videos are 10-15 minutes in duration and are intended to teach behavioral principles for losing weight, healthy eating, and exercise.
  Arms: Automated online program + coaching; Automated online program only
Behavioral: Individual coaching — Participants will receive monthly, one-on-one coaching sessions (12 in total) throughout the 12-month intervention period. Coaching sessions will be conducted via videoconference and the initial coaching session will be approximately 30 minutes and all remaining sessions will be approximately 15 minutes. The structure of the coaching sessions will be similar across participants, but the content will be tailored to the individual. Coaches will use goal setting, problem solving, and motivational interviewing to help facilitate adherence and achievement of weight loss program goals.
  Arms: Automated online program + coaching; Group videoconference program + coaching
Behavioral: Group-based, videoconference-delivered weight loss — Participants receiving this program will be instructed to attend interactive group videoconference sessions (60 minutes each) focused on behavioral strategies for changing diet and exercise to promote weight loss. Classes will be weekly during months 1-3, twice per month during months 4-6, and monthly during months 7-12. These classes are designed to allow participants to interact with, support, and learn from one another. Participants are also given a daily calorie intake goal of 1200-1800 kcal/day based upon their starting weight and a moderate-intensity aerobic exercise (e.g., walking) goal which progresses to 250 min/week. They are instructed to self-monitor body weight, calorie intake, and exercise minutes daily over 12 months, and are provided with a smart scale for electronic transmission of weight data. Semi-automated, personalized feedback, based on self-monitoring data, is provided by the group instructor at the same frequency as group sessions are held.
  Arms: Group videoconference program + coaching; Group videoconference program only

SUMMARY:
The purpose of this trial is to compare two delivery formats for weight loss (automated online program vs. group-based videoconference program) and to examine the added effect of individual coaching (vs. no coaching) for individuals with overweight or obesity. All participants enrolled in this study will receive a 12-month behavioral weight loss program (varying in delivery format and individual support), and will be provided with weight loss, calorie intake, and exercise goals. Assessments will occur at baseline, 6 (mid-treatment), 12 (post-treatment), and 18 months (following 6 months of no intervention). We will also seek to determine which combination of intervention approaches works best for whom and develop algorithms which can be used to refer patients into remote programs in clinical settings or future trials.

DETAILED DESCRIPTION:
Participants will be randomized at baseline to one of four weight loss intervention conditions: 1) automated program + coaching, 2) automated program + no coaching, 3) group videoconference program + coaching, and 4) group videoconference program + no coaching. All participants will be provided with weekly goals, instructed to self-monitor diet, exercise, and weight daily, and provided with feedback based upon these data. Those receiving the online program will also be instructed to view video lessons (24 in total, 10-15 min each) which focus on behavioral strategies for changing diet and exercise. Individuals randomized to the videoconference program will participate in 24 group sessions (1 hour each) designed to mimic in-person treatment and allow for participant interaction via large and small group discussions. The content across conditions will be similar and the lessons will be provided weekly during months 1-3, twice per month during months 4-6, and monthly during months 7-12. Those receiving coaching will have individual, monthly meetings with a coach via videoconference (~15 min each). Coaching sessions will focus on individual barriers, problem solving, goal setting, and fostering support and accountability.

The primary aim of this study is to examine the effects of delivery format (automated online vs. videoconference) and coaching (individualized vs. none) on weight loss at 12 months. Secondary aims will examine the effects of delivery format and coaching on intervention engagement (e.g., frequency of self-monitoring), psychosocial outcomes (e.g., perceived support, self-efficacy, and motivation), 18-month weight loss, and the cost per kilogram of weight loss (to examine whether the addition of human support is cost-effective). Two algorithms will also be developed to predict which treatment type should be recommended to whom, using only baseline characteristics: 1) a 'widely-applicable' algorithm which will use metrics common to electronic medical records (sex, BMI, age, race, ethnicity), and 2) a 'more comprehensive' algorithm which will further include additional baseline characteristics (e.g., education, household income, health literacy, group preference, etc).

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index between 25-45 kg/m2
* Daily, home Internet access

Exclusion Criteria:

* Currently pregnant, planning to become pregnant within the next 18 months, or pregnant within the past 6 months
* Current or recent enrollment (<2 years) in a weight loss program
* Presence of any medical condition for which exercise, weight loss, or dietary restriction is contraindicated
* Recent weight loss (≥10 pounds within the past 6 months)
* Currently taking weight loss medications or history of bariatric surgery
* Inability to walk 2 blocks without stopping
* Non-English speaking
* A member of one's household is participating in the study
* History of anorexia or bulimia nervosa

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 490 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2028-04-27 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Percent weight change | 12 months
  Weight change will be assessed via smart scales using weight at baseline and 12 months and calculated as follows: ([12-month weight minus baseline weight] / baseline weight * 100).
Change in perceived support | 12 months
  Perceived support will be measured via the Important Others Questionnaire. Scores on this questionnaire range from 12 to 84 with higher scores indicating a greater perception of support from important others. Change in perceived support will be calculated as follows: 12-month perceived support minus baseline perceived support.

SECONDARY OUTCOMES:
Cost per kilogram of weight loss | 12 months
  The cost per participant to deliver the intervention will be calculated and divided by the average weight change (in kilograms) from baseline to 12 months.
Percent weight change | 18 months
  Weight change will be assessed via smart scales using weight at baseline and 18 months and calculated as follows ([18 month weight minus baseline weight] / baseline weight * 100).
Frequency of self-monitoring weight | 12 months
  The number of days that a participant stepped on the scale over the 12-month intervention period will be calculated.
Self-monitoring of calorie intake | 12 months
  The number of days that a participant reported their calorie intake over the 12-month intervention period will be calculated.
Change in self-efficacy for diet | 12 months
  Self-efficacy for diet will be measured via the Weight Efficacy Lifestyle Questionnaire. Scores range from 0 to 80, with higher scores indicating greater self-efficacy. Change in self-efficacy for diet will be calculated as 12-month score minus the baseline score.
Self-efficacy for exercise | 12 months
  Self-efficacy for exercise will be measured via the Self-Efficacy for Exercise Scale. Scores range from 0 to 90 with higher scores indicating greater self-efficacy. Change in self-efficacy for exercise will be calculated as the 12-month score minus the baseline score.
Change in autonmous motivation | 12 months
  Autonomous motivation will be measured via the Treatment Self-Regulation Questionnaire for Weight Management (autonomous motivation subscale). Scores range from 6 to 42 and higher scores indicate more autonomous motivation. Change in motivation will be calculated as the 12-month score minus the baseline score.
Change in controlled motivation | 12 months
  Controlled motivation will be measured via the Treatment Self-Regulation Questionnaire for Weight Management (controlled motivation subscale). Scores range from 6 to 42 and higher scores indicate more controlled motivation. Change in motivation will be calculated as the 12-month score minus the baseline score.

CONTACTS AND LOCATIONS:
Locations (1):
- The Miriam Hospital's Weight Control and Diabetes Research Center, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF